CLINICAL TRIAL: NCT07348549
Title: THE EFFECT OF BREAST CANCER EDUCATION CONDUCTED WITH THE GAGNE LEARNING MODEL ON KNOWLEDGE, ATTITUDES TOWARDS LEARNING, AND CRITICAL THINKING SKILLS OF NURSING STUDENTS
Brief Title: Gagne Learning Model in Nursing Education
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Dilek Erden, Principal Investigator, Dr. Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DERDEN-3
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Nursing Education; Learning Process in Nursing Graduation; Learning Techniques
Keywords: Gagne learning model; Nursing educaiton; Nursing student; Critical thinking; Attitude towards learning

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- Gagne Learning Model (Experimental): Group receiving training with the Gagne learning model
  Interventions: Other: Gagne Learning group
- Control Group- Traditional Learning Model (Placebo Comparator): Groups receiving education through the traditional learning model
  Interventions: Other: Control group- Traditional learning model

INTERVENTIONS:
Other: Gagne Learning group — Group receiving training with the Gagne learning model
  Arms: Intervention group- Gagne Learning Model
Other: Control group- Traditional learning model — Groups receiving education through the traditional learning model
  Arms: Control Group- Traditional Learning Model

SUMMARY:
This study aims to examine the effect of breast cancer education, conducted using the Gagne learning model, on nursing students' knowledge, attitudes towards learning, and critical thinking skills.

DETAILED DESCRIPTION:
The study is a randomized controlled trial with experimental and control groups. The study implements an educational program based on Gagne's learning model and a traditional learning model. Data are collected using a comprehensive breast cancer knowledge test, an attitude scale toward learning, a critical thinking skills questionnaire, and a self-breast examination teaching skills form.

ELIGIBILITY:
Inclusion Criteria:

* Third-year students who had taken courses in fundamentals of nursing, internal medicine nursing, physiology, pathology, and computer science, but had not taken oncology nursing, were included in the study as volunteers.

Exclusion Criteria:

* Students who were not in their third year of study, did not take one of the following courses: fundamentals of nursing, internal medicine nursing, physiology, pathology, computer science, those who had taken the oncology nursing course, and those who did not volunteer to participate in the research were excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Breast Cancer Knowledge Test | 4 weeks
  The comprehensive beast cancer knowledge test consists of 20 general knowledge questions. The scale is answered using a True-False format. There are 8 true and 12 false statements. The comprehensive breast cancer knowledge test comprises two dimensions: general knowledge and treatability. Questions 1 through 12 cover general knowledge about breast cancer, while questions 13 through 20 concern the treatability of breast cancer.

SECONDARY OUTCOMES:
Attitudes Towards Learning Scale | 4 weeks
  The attitude towards learning scale consists of a total of 34 items. The scale comprises sub-dimensions of effort toward learning, valuing learning, and avoidance of learning. Of these items, 25 are positive and 9 are negative. The scale is rated on a 5-point Likert scale, with options being "Strongly Agree", "Largely Agree", "Partially Agree", "Disagree", and "Strongly Disagree". The highest possible attitude score is 170 and the lowest is 34.

OTHER OUTCOMES:
Critical Thinking Skills Questionnaire | 4 weeks
  The scale is the "Critical Thinking Skills Questionnaire". Consisting of 22 items on a 5-point Likert scale, the critical thinking skills questionnaire assigns scores to participants for each question on a scale of 1 (Strongly Disagree), 2 (Disagree), 3 (Undecided), 4 (Agree), and 5 (Strongly Agree).
Self-Breast Examination Teaching Skill Form | 4 weeks
  The "Self-Breast Examination Teaching Skill Form," is included in the Birth and Women's Health Practice Guide for Nurses and Midwives. The form, which uses a 3-point likert scale, consists of 22 skill stages. The form includes application columns (1, 2, 3) depending on whether or not the successful behavior is demonstrated. The form consists of two parts: process and product. In the evaluation process, each item is given one point, with the process dimension receiving a total of 22 points and the product dimension receiving 5 points, for a total of 27 points.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK ERDEN, Principal Investigator — Namik Kemal University
Locations (1):
- Tekirdag Namık Kemal University, Tekirdağ, Namık Kemal Street, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share it with researchers who request it for reasonable reasons.

REFERENCES:
- [Background] Tang, W. L., Tsai, J. T., & Huang, C. Y. (2020). Inheritance coding with Gagné-based learning hierarchy approach to developing mathematics skills assessment systems. Applied Sciences, 10(4), 1465.